CLINICAL TRIAL: NCT00749593
Title: Cross-Sectional Multi-Centre Study of UK Adults With Congenital Adrenal Hyperplasia.
Brief Title: Study of UK Adults With Congenital Adrenal Hyperplasia.
Acronym: CaHASE
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Society for Endocrinology (Other); The Clinical Endocrinology Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: STH13503; MREC 04/07/013
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; Quality of Life; Genotype; Metabolic outcomes
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CaHASE 1: Adults with CAH

SUMMARY:
Congenital Adrenal Hyperplasia (CAH) is one of the commonest inherited diseases, affecting 1:14,200 live births. It is the result of a genetic defect in one of the enzymes (in most cases 21-hydroxylase) required for cortisol biosynthesis, leading to reduced levels of cortisol and aldosterone, increased ACTH concentrations and consequently increased adrenal androgen production. Patients suffer from problems with growth and development and as adults patients may have problems with fertility, virilisation in women, testicular masses in men and both men and women have an impaired quality of life. Patients have to take life-long therapy. Despite its frequency knowledge surrounding the management of adults with CAH remains fairly limited. There has been a lot of work describing the management of children with CAH but to date there is no consensus on how to manage adults. To address this issue a number of adult endocrinologists in the UK under the auspices of the Society for Endocrinology have established a country wide study (CaHASE) to undertake research in order to set standards of care for adult patients with CAH.

In CAH the severity of the symptoms experienced by affected individuals varies depending on the mutation and the genetic background of the individual. The ability to tailor CAH therapy on an individual basis, as determined by the severity of the underlying defect and an understanding of the likely natural history of the disease, is a key goal in clinical management. Correlation of phenotype (clinical status) and genotype (the underlying 21 hydroxylase gene mutation) will facilitate stratification of severity and provide an important contribution to the debate on potential mechanisms of individualised therapy. For instance it may become clear that certain CAH genotypes are associated with specific long term outcomes. In time, this could lead to suggesting different treatment strategies in certain groups. Moreover, genotype data are important if we are to address the relative contribution of environment (e.g. treatment) vs. genetics on long term outcomes.

This multi-centre study aims to:

1. - Investigate the medical health of adults with congenital adrenal hyperplasia.
2. - Investigate the relationship between the genotype of the patient and the phenotype.
3. - Investigate the quality of life of adults with congenital adrenal hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Clinical and genetic diagnosis of congenital adrenal hyperplasia

Exclusion Criteria:

* Pregnant females
* Under 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK Adults with Congenital Adrenal Hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-08; Primary Completion 2007-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The anthropometric, metabolic, endocrine and quality of life variables of adults with congenital adrenal Hyperplasia will be compared to reference ranges for the normal population. | End of Study

SECONDARY OUTCOMES:
To identify areas where further research is required and to inform on the day to day management of adults with CAH | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Richard JM Ross, MD, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, United Kingdom

REFERENCES:
- [Derived] Han TS, Conway GS, Willis DS, Krone N, Rees DA, Stimson RH, Arlt W, Walker BR, Ross RJ; United Kingdom Congenital Adrenal Hyperplasia Adult Study Executive (CaHASE). Relationship between final height and health outcomes in adults with congenital adrenal hyperplasia: United Kingdom congenital adrenal hyperplasia adult study executive (CaHASE). J Clin Endocrinol Metab. 2014 Aug;99(8):E1547-55. doi: 10.1210/jc.2014-1486. Epub 2014 May 30. PMID 24878054
- [Derived] Krone N, Rose IT, Willis DS, Hodson J, Wild SH, Doherty EJ, Hahner S, Parajes S, Stimson RH, Han TS, Carroll PV, Conway GS, Walker BR, MacDonald F, Ross RJ, Arlt W; United Kingdom Congenital adrenal Hyperplasia Adult Study Executive (CaHASE). Genotype-phenotype correlation in 153 adult patients with congenital adrenal hyperplasia due to 21-hydroxylase deficiency: analysis of the United Kingdom Congenital adrenal Hyperplasia Adult Study Executive (CaHASE) cohort. J Clin Endocrinol Metab. 2013 Feb;98(2):E346-54. doi: 10.1210/jc.2012-3343. Epub 2013 Jan 21. PMID 23337727
- [Derived] Arlt W, Willis DS, Wild SH, Krone N, Doherty EJ, Hahner S, Han TS, Carroll PV, Conway GS, Rees DA, Stimson RH, Walker BR, Connell JM, Ross RJ; United Kingdom Congenital Adrenal Hyperplasia Adult Study Executive (CaHASE). Health status of adults with congenital adrenal hyperplasia: a cohort study of 203 patients. J Clin Endocrinol Metab. 2010 Nov;95(11):5110-21. doi: 10.1210/jc.2010-0917. Epub 2010 Aug 18. PMID 20719839